CLINICAL TRIAL: NCT04046094
Title: IV Vitamin C With Chemotherapy for Cisplatin Ineligible Bladder Cancer Patients: A Forgotten Group
Brief Title: Intravenous (IV) Vitamin C With Chemotherapy for Cisplatin Ineligible Bladder Cancer Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, John Taylor, Professor, Director of Basic Urologic Research, Co-Leader of D3ET, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2019-IVC_CarboGem; UL1TR002366 (NIH)
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer
Keywords: Intravenous (IV) Ascorbic Acid (Vitamin C)
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: To assess pathologic downstaging rate in MIBC cisplatinineligible patients when IVC is added to a gemcitabine/carboplatin NAC regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IV Ascorbic Acid (Experimental): IV Ascorbic Acid 25 grams (g) infused 2 times a week for 4 weeks
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — Ascorbic Acid Intravenous
  Other Names: Vitamin C

SUMMARY:
Bladder cancer is a common disease with high rates of mortality, especially at advanced stages. Neo-adjuvant cisplatin-based chemotherapy (NAC) followed by radical cystectomy is considered standard of care for patients with muscle invasive disease, as NAC improves surgical outcomes in these patients. However, some patients are ineligible for cisplatin-based chemotherapy due to other medical issues. Although a combination of carboplatin and gemcitabine has been used with limited success, most patients proceed directly to cystectomy without realizing the potential survival benefit afforded by NAC. Intravenous ascorbate (vitamin C) administration (IVC) has been shown to improve both carboplatin and gemcitabine-based therapy in other models. This trial will add IVC to gemcitabine/carboplatin chemotherapy to evaluate whether co-treatment will increase therapeutic efficacy.

DETAILED DESCRIPTION:
see protocol

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status = 0 -- 2
* Cisplatin-ineligible, muscle invasive bladder cancer
* Adequate organ and marrow functions
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use protocol specified forms of birth control

Exclusion Criteria:

* Patient simultaneously enrolled in any therapeutic clinical trial
* Current or anticipated use of other investigational agents while participating in this study
* Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast feeding. There is a potential for congenital abnormalities and for this regimen to harm breast feeding infants
* Histology of pure adenocarcinoma, pure squamous cell carcinoma, or pure small cell carcinoma in the TURBT sample
* Prior systemic chemotherapy (prior intravesical therapy is allowed) and/ or prior radiation therapy to the urinary bladder
* Uncontrolled intercurrent illness
* Current consumption of tobacco products
* History of glucose-6-phosphate dehydrogenase (G6PD) deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2026-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Taylor, MD MS, Principal Investigator — The University of Kansas
Locations (3):
- United States (3):
  - The University of Kansas Cancer Center (KUCC), Fairway, Kansas
  - The University of Kansas Medical Center, Kansas City, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Ascorbic Acid
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IV Ascorbic Acid
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Post Treatment Pathological Staging
Description: Post treatment specimen pathology results evaluated per the WHO TNM staging system. The staging system is a qualitative assessment based on the results of the physical exam, biopsy, imaging tests, and the results of surgery. The earliest stage cancers are called stage 0 (or carcinoma in situ), and then range from stages I (1) through IV (4). As a rule, the lower the number, the less the cancer has spread. A higher number, such as stage IV, means a more advanced cancer.
Time Frame: 6 weeks after first IVC infusion at radical cystectomy
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ascorbic Acid
Number analyzed (Participants) | 12
Participants
  Stage 0 | 3
  Stage I | 2
  Stage II | 1
  Stage III | 4
  Stage IV | 2

2. Secondary Outcome: Overall Change in Patient-reported Quality of Life Outcomes
Description: Scores evaluated per Functional Assessment of Cancer Therapy - Bladder (FACT-Bl) version 4 - quality of life (QOL) questionnaire scores:
  * FACT-Bl total score range is 0-156, derived by the sum of the sub-scales. Higher scores indicate better QOL.
  * FACT-Bl includes five sub-scales:
    * Physical Well-being (PWB), score range of 0-28
    * Social/Family Well-being (SWB), score range of 0-28
    * Emotional Well-being (EWB), score range of 0-24
    * Functional Well-being (FWB), score range of 0-28
    * Bladder Cancer Subscale (BlCS), score range of 0-48
  * Note: Negatively stated items are reversed by subtracting the response from "4".
Time Frame: Baseline, End of Treatment (completion of neoadjuvant therapy, Day 28), Post-surgery (6 weeks post-operative)
Reporting Status: Not Posted, anticipated posting 2025-08

3. Secondary Outcome: Disease Free Survival Rate (DFS) Among Participants
Description: DFS will be defined as time from cystectomy to disease recurrence or death resulting from disease. DFS represents time from random assignment to cancer recurrence or death from any cause. Patients alive without disease progression at the time of analysis were censored at the date of last disease assessment.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2025-08

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | IV Ascorbic Acid
All-Cause Mortality (participants affected / at risk) | 4/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Ascorbic Acid (N=12)
Ileus (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT04046094/Prot_SAP_000.pdf